CLINICAL TRIAL: NCT01357486
Title: Phase II Randomized Trial Evaluating the Administration of Sorafenib or Pravastatin or Association Sorafenib-pravastatin or Best Supportive Care for the Palliative Treatment of Hepatocellular Carcinoma in Patient With CHILD B Cirrhosis
Brief Title: Palliative Treatment of Hepatocellular Carcinoma in Patient With CHILD B Cirrhosis
Acronym: PRODIGE 21
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Federation Francophone de Cancerologie Digestive (Other); UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2010/22
Record Dates: First submitted 2011-05-13; First posted 2011-05-20 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Hepatocellular Carcinoma; CHILD B
Keywords: Hepatocellular Carcinoma; CHILD B; palliative management; Sorafenib; Pravastatin
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Experimental): patients receiving sorafenib 400 mg - twice a day
  Interventions: Drug: sorafenib
- B (Experimental): patients receiving pravastatin 40 mg - once a day
  Interventions: Drug: Pravastatin
- C (Experimental): patients receiving sorafenib 400 mg (twice a day) and pravastatin 40 mg (once a day)
  Interventions: Drug: Sorafenib + Pravastatin
- D (Other): patients receiving best supportive care
  Interventions: Other: patients receiving best supportive care

INTERVENTIONS:
Drug: sorafenib — patients receiving sorafenib 400 mg - twice a day
  Arms: A
Drug: Pravastatin — patients receiving pravastatin 40 mg - once a day
  Arms: B
Drug: Sorafenib + Pravastatin — patients receiving sorafenib 400 mg (twice a day) and pravastatin 40 mg (once a day)
  Arms: C
Other: patients receiving best supportive care — palliative management
  Arms: D

SUMMARY:
The incidence of Hepatocellular Carcinoma (HCC) is currently increasing in Europe and in France and about 2 / 3 of patients, are not eligible for curative treatment at the time of diagnosis. The palliative management of patients with advanced and symptomatic disease is complex and requires treatment combining anti-tumor activity and safety in patients with impaired liver functions. Sorafenib is the standard of care in a palliative setting, but the benefit of sorafenib in patient with altered liver function is uncertain. The aim of this trial is to study the interest of sorafenib in patients with HCC and impaired liver function compared to pravastatin (a drug with anti-tumoral activity in HCC) or to the combination sorafenib/pravastatin or to best supportive care (usually used in these patients).

DETAILED DESCRIPTION:
The incidence of Hepatocellular Carcinoma (HCC) is currently increasing in Europe and in France. It almost always occurs on liver disease and in 80 to 90% of cases, at least in France, on liver with cirrhosis. If curative treatment may be proposed for some "small" HCC (transplantation, resection, percutaneous destruction), about 2 / 3 of patients, which represents nearly 4,000 new cases per year in France, are not eligible for such treatment. The palliative management of patients with advanced and symptomatic disease is complex and requires treatment combining anti-tumor activity and safety in patients with impaired liver functions. Indeed, in most cases the palliative treatment of HCC is applied to patients with altered liver function (stage B of the Child-Pugh classification).

To date, the proposed treatment in France for such patients is based on best supportive care.

The objective of this study is to assess the interest in this situation of 2 molecules - taken alone or in combination:

* Sorafenib, the reference in the palliative treatment of advanced hepatocellular carcinoma (Stage C of the BCLC classification). Yet the safety and efficacy of sorafenib in patients with altered liver function (CHILD B) are not clearly defined and its use remains discouraged by French recommendations in these patients.
* Pravastatin whose interest in the palliative treatment of HCC was suggested by several phase II studies with a good safety profile in cirrhotic patients.

In this French multicenter open randomized study, 160 patients will be included in 4 arms (40/arms): sorafenib, pravastatin, pravastatin + sorafenib, and supportive care.

The aim of this phase II multicenter study is to select the two best arms for further Phase III study in order to identify a reference treatment in this palliative situation.

ELIGIBILITY:
Inclusion Criteria:

- Male and female subjects > 18 years age

- Hepatocellular carcinoma histologically diagnosed or in case of inability to perform a histology by non invasive radiological criteria in presence of known cirrhosis: (i) Hepatic lesion measuring between 1 and 2 cm in diameter : CT-scan + MRI (eventually an Ultrasound contrast) : HCC diagnosed with contrast uptake in the arterial phase and rapid wash out in the venous /late phase on two imaging techniques.

(ii)Hepatic lesion with a diameter > 2 cm : CT-scan or MRI +alpha fetoprotein : HCC diagnosed with contrast uptake in the arterial phase and a rapid wash out in the venous /late phase or a alpha fetoprotein > 200µg/L

* Patient not eligible for curative treatment (transplantation, resection, destruction or percutaneous chemo-embolization) or HCC still evolving after failure of a specific treatment
* Score CHILD B
* ECOG performance status 0/1/2
* Score BCLC B or C
* Adequate haematologic function with haemoglobin > 8 g/dl, platelet count > 50000x 109/L, absolute neutrophil count > 1000 / mm3
* Creatinine < 2 times the upper limit of normal
* Written informed consent

Exclusion Criteria:

* Any condition that is unstable or could jeopardize the safety of the subject and their compliance in the study
* Pregnancy
* Myocardial infarction less than 6 months, uncontrolled hypertension, congestive heart failure(NYHA class > 2) , anti- arrhythmic treatment other than beta-blockers or digoxin
* Digestive bleeding within 30 days before inclusion
* Hepatic transplantation
* Patients receiving or having received a statine for less than 6 months before HCC diagnostic
* Prior use of sorafenib
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Previous or concurrent cancer, except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumor. Any cancer curatively treated > 5 years prior to entry is permitted
* Known or suspected history of allergy to sorafenib or pravastatin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-11-14 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Time to radiologic progression | Every 4 weeks (CT-scan or MRI) until progression of HCC or date of last news (for patients alive or dead without progression)

SECONDARY OUTCOMES:
Overall survival | End of the study (estimated date August 2012)
Survival without progression | Every 4 weeks (CT-scan or MRI) until progression of HCC or date of last news (for patients alive or dead without progression)
Time to treatment failure | every 4 weeks (CT-scan or MRI) until clinical or radiological progression of HCC or date of last news (for patients alive or dead without progression)
Objective response rate at four months | Radiological evaluation at 4 months
Number and description of AE for toxicity and SAE | Clinical evaluation every month
Quality of life | Clinical evaluation every month

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Frédéric BLANC, MD-PhD, Principal Investigator — University Hospital, Bordeaux
Locations (35):
- France (35):
  - CH d'Abbeville, Abbeville
  - CH Pays d'Aix, Aix-en-Provence
  - CH d'Auxerre, Auxerre
  - CH de la Côte Basque, Bayonne
  - CH de Béziers, Béziers
  - AP-HP- Hôpital Jean-Verdier, Bondy
  - CHU de Bordeaux, Bordeaux
  - CH Duchenne, Boulogne-sur-Mer
  - AP-HP Hôpital Henri Mondor, Créteil
  - CHU Le Bocage, Dijon
  - CH Départemental Vendée, La Roche-sur-Yon
  - CH Le Mans, Le Mans
  - CH de Bretagne Sud, Lorient
  - Hôpital privé Jean Mermoz, Lyon
  - AP-HM Hôpital de la Timone, Marseille
  - CH de Meaux, Meaux
  - CH Mont de Marsan, Mont-de-Marsan
  - CHU de Nancy Hôpital Brabois, Nancy
  - CHU de Nantes Hôpital de l'Hotel Dieu, Nantes
  - CHU Nîmes, Nîmes
  - CHR d'Orléans - Hôpital La Source, Orléans
  - Groupe Hospitalier Paris Saint Joseph, Paris
  - CH Perpignan, Perpignan
  - CHU de Bordeaux, Hôpital du Haut Lévèque, Pessac
  - CH de la Région d'Annecy, Pringy
  - Centre Eugène Marquis, Rennes
  - Clinique Mathilde, Rouen
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - Centre René Gauducheau CLCC Nantes Atlantique, Saint-Herblain
  - CH Gaston Ramon, Sens
  - CH Saint-Malo, St-Malo
  - Centre Régional de Lutte contre le Cancer Centre Paul Strauss, Strasbourg
  - Hôpitaux Universitaires de Strasbourg Hôpital civil, Strasbourg
  - Hôpitaux Universitaires de Strasbourg, Hôpital Hautepierre, Strasbourg
  - CHRU de Tours, Tours

REFERENCES:
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Taras D, Blanc JF, Rullier A, Dugot-Senant N, Laurendeau I, Vidaud M, Rosenbaum J. Pravastatin reduces lung metastasis of rat hepatocellular carcinoma via a coordinated decrease of MMP expression and activity. J Hepatol. 2007 Jan;46(1):69-76. doi: 10.1016/j.jhep.2006.06.015. Epub 2006 Jul 28. PMID 16935385
- [Background] Kawata S, Yamasaki E, Nagase T, Inui Y, Ito N, Matsuda Y, Inada M, Tamura S, Noda S, Imai Y, Matsuzawa Y. Effect of pravastatin on survival in patients with advanced hepatocellular carcinoma. A randomized controlled trial. Br J Cancer. 2001 Apr 6;84(7):886-91. doi: 10.1054/bjoc.2000.1716. PMID 11286466
- [Background] Lersch C, Schmelz R, Erdmann J, Hollweck R, Schulte-Frohlinde E, Eckel F, Nader M, Schusdziarra V. Treatment of HCC with pravastatin, octreotide, or gemcitabine--a critical evaluation. Hepatogastroenterology. 2004 Jul-Aug;51(58):1099-103. PMID 15239254
- [Background] Cohen DE, Anania FA, Chalasani N; National Lipid Association Statin Safety Task Force Liver Expert Panel. An assessment of statin safety by hepatologists. Am J Cardiol. 2006 Apr 17;97(8A):77C-81C. doi: 10.1016/j.amjcard.2005.12.014. Epub 2006 Feb 3. PMID 16581333
- [Background] Llovet JM, Di Bisceglie AM, Bruix J, Kramer BS, Lencioni R, Zhu AX, Sherman M, Schwartz M, Lotze M, Talwalkar J, Gores GJ; Panel of Experts in HCC-Design Clinical Trials. Design and endpoints of clinical trials in hepatocellular carcinoma. J Natl Cancer Inst. 2008 May 21;100(10):698-711. doi: 10.1093/jnci/djn134. Epub 2008 May 13. PMID 18477802
- [Derived] Blanc JF, Khemissa F, Bronowicki JP, Monterymard C, Perarnau JM, Bourgeois V, Obled S, Abdelghani MB, Mabile-Archambeaud I, Faroux R, Seitz JF, Locher C, Senellart H, Villing AL, Audemar F, Costentin C, Deplanque G, Manfredi S, Edeline J; PRODIGE 21 collaborators. Phase 2 trial comparing sorafenib, pravastatin, their combination or supportive care in HCC with Child-Pugh B cirrhosis. Hepatol Int. 2021 Feb;15(1):93-104. doi: 10.1007/s12072-020-10120-3. Epub 2021 Jan 9. PMID 33420951